CLINICAL TRIAL: NCT05619991
Title: Effect of Short Film Video and Video-Based Education on Fear, Pain, and Satisfaction of Children Undergoing Day Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, Gamze BOZKUL, Research asistant, Tarsus University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TU-BOZKUL-001
Record Dates: First submitted 2022-11-09; First posted 2022-11-17 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Day Surgery; Fear; Pain; Satisfaction; CHİLDREN
MeSH Terms: conditions — Pain; Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group watching video (Experimental): For the Educational Video, a scenario appropriate for the age group, about the preparation for the surgery, the operating room environment and the post-operative process will be created by the researchers. Expert opinion will be taken for the suitability of the scenario.
  Interventions: Other: Group watching video
- Scheduled training group (Other): For the Planned Education, a power point presentation will be prepared by the researchers, appropriate for the age group, about the preparation for the surgery, the operating room environment and the post-operative process, and the patients will be trained before the surgery.
  Interventions: Other: Scheduled training group
- Control group (No Intervention): Before the operation, the fear and vital signs of the children in the sample will be evaluated. In the postoperative period, the pain, fear and vital signs of the children in the control group will be recorded and a questionnaire examining the satisfaction status will be applied.

INTERVENTIONS:
Other: Group watching video — The video will include preparation for the surgery, the operating room environment and the post-operative process.
  Arms: Group watching video
Other: Scheduled training group — The scheduled training will include preparation for the surgery, the operating room environment and the post-operative process.
  Arms: Scheduled training group

SUMMARY:
It is aimed to investigate the effect of introducing the operating room environment with an informative video to pediatric patients aged 7-12 in the preoperative period in day surgery on pain, fear, and patient and parent satisfaction. In line with this purpose, an answer was sought to the question "How did the different education programs given to children who will undergo day surgery have an effect on fear, pain and satisfaction?" It will be conducted in a single center, parallel group, randomized controlled experimental design. The research will be carried out between December 2022 and October 2023 and it is planned to continue for 12 months. The population of the research will be children between the ages of 7-12 who will undergo a day surgery at Tarsus State Hospital, and the sample will be 90 children who meet the criteria for inclusion in the research. Considering that there may be case losses, a total of 90 children (1st experimental group [watched video training]:30 children, 2nd experimental group [provided planned training]: 30 children, control group: 30 children) will be included in the sample group. In the collection of research data; Introductory Information Form, Numerical Pain Scale, Child Fear Scale, Vital Signs Follow-up Form (Appendix 4) will be used. The application will be started after the approval of the ethics committee and the written permission of the institution for the research. Statistical package program (SPSS 20) will be used in the analysis of the research data.

DETAILED DESCRIPTION:
In this study, it is aimed to investigate the effect of introducing the operating room environment with an informative video to pediatric patients aged 7-12 in the preoperative period in day surgery on pain, fear, and patient and parent satisfaction. It will be conducted in a single center, parallel group, randomized controlled experimental design. Randomization will be provided by randomly and evenly distributing the patients who meet the sample selection criteria into 3 groups (1st experimental group, 2nd experimental group and 3rd group control group) through a program in the computer environment. (http://www1.assumption.edu/users/avadum/applets/RandAssign/GroupGen.html). The application will be started after the approval of the ethics committee and the written permission of the institution for the research.

Stage 1: The information content to be included in the video will be determined by the researchers, taking the opinions of the experts on the subject, appropriate for the level of the child in the 7-12 age group, for daily surgical intervention (about preparation for surgery, the operating room environment and the post-operative process), and video content will be created. .

Stage 2: In line with the suggestions from researchers and experts, an informative video will be prepared for day surgery (preparation for surgery, operating room environment and the post-operative process) appropriate for the level of the child in the 7-12 age group.

Stage 3: A pilot study will be conducted with 10 children in order to evaluate the data collection forms to be used before the research and the suitability of video education for children.

Stage 4: The children in the sample group and their parents will be informed about the method followed in practice and the research, and verbal and written consent will be obtained.

Stage 5: The introductory information form in the research will be applied to the children in the sample group.

Stage 6: Patients who meet the sample selection criteria will be randomly and equally distributed into 2 groups (1st experimental group, 2nd experimental control group and 3rd group control group) through a program in the computer environment, and randomization will be achieved.

(http://www1.assumption.edu/users/avadum/applets/RandAssign/GroupGen.html). Stage 7: The children in the experimental group will be shown an informative video prepared.

Stage 8: Before the operation, the fear and vital signs of the children in the sample will be evaluated.

Stage 9: In the postoperative period, pain, fear, vital signs of the children in the experimental and control groups will be recorded and a questionnaire examining the satisfaction status will be applied.

Written approval from Mersin University Clinical Research Ethics Committee, written institutional permission from Tarsus State Hospital, and informed written consent from parents and children will be obtained before the research data begins to be collected. The population of the research will be children between the ages of 7-12 who will undergo outpatient surgery in Tarsus State Hospital, and the sample will be 90 children who meet the criteria for inclusion in the research. Randomization was made between the control and treatment groups by stratification in terms of children, gender and age variables. According to this randomization method, homogeneity is achieved between the groups (Kanik, Taşdelen, & Erdoǧan, 2011). The sample of the research was determined by G power power analysis by consulting a statistician. In the study, power analysis was performed to determine the number of people to work in two groups. The power of the test was calculated with the G*Power 3.1 program. For the power of the work to exceed 80%; 5% significance level and 0.80 effect level; It is necessary to reach a total of 78 people, with a minimum of 26 people in the groups (t=2009; Effect size d=0.80). Considering that there may be case losses, a total of 90 children (1st experimental group [watched video training]:30 children, 2nd experimental group [provided planned training]: 30 children, control group: 30 children) will be included in the sample group.

ELIGIBILITY:
Inclusion Criteria:

* To be 7 and 12 years old
* Having day surgery
* Not having undergone previous surgery
* Not have a chronic disease
* No communication, mental or neurological problems
* Volunteering to participate in the study

Exclusion Criteria:

* Not be in the 7-12 age range
* Not to have day surgery
* Having had previous surgery
* have a chronic illness
* Having another chronic illness
* Have a communication, mental, or neurological problem
* Not willing to participate in the study

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-22 (Actual)

PRIMARY OUTCOMES:
Introductory Information Form | 1 day
  Introductory Information Form, which was created by the researcher in line with the knowledge of the literature, consists of questions about the child's age, gender, educational status, and characteristics of the procedure (Baghele et al., 2019; Eijlers et al., 2019; Yaz & Yılmaz, 2021).
Child Fear Scale | 1 day
  Child Fear Scale, McKinley et al. (2003) as "The Faces Anxiety Scale" for adult patients. The same scale was adapted for pediatric patients as "Children's Fear Scale" by McMurtry et al. (2011). This Scale includes 5 different facial expressions. This scale is scored between 0 and 4, and it is stated to be a reliable and valid measurement tool in the evaluation of fear.
Numerical Pain Scale | 1 day
  Numerical Pain Scale, this method for determining the severity of pain, aims to explain the patient's pain in numbers. Absence of pain (0) is evaluated as unbearable pain (10) on numerical scales.
The Vital Signs Follow-up Form | 1 day
  The Vital Signs Follow-up Form was prepared to record the vital signs of children measured before and immediately after the procedure, such as heart rate, blood pressure, saturation value and respiration.
The Child Satisfaction Scale | 1 day
  The Child Satisfaction Scale was developed by researchers in a way that children can easily understand (Çelik, 2020). The numbers between 0 and 10, which the children would indicate by circling the point corresponding to their satisfaction with the education provided, were placed on a horizontal line. On the scale, 0 points means "not at all satisfied" and 10 points means "extremely satisfied". In addition, images reflecting the degree of satisfaction have been added to the places where the scores are located. In the study, it is planned to be applied to all groups after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Atiye Karakul, Assoc. Prof., Study Director — Tarsus University; Duygu Sönmez Düzkaya, Assoc. Prof., Principal Investigator — Tarsus University; Şahika Dilşen, Uzm. Dr., Principal Investigator — TARSUS STATE HOSPİTAL; Gamze Bozkul, Res. Ass., Principal Investigator — Tarsus University
Locations (2):
- Turkey (Türkiye) (2):
  - Gamze Bozkul, Mersin
  - Tarsus University, Mersin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bartik K, Toruner EK. Effectiveness of a Preoperative Preparation Program on Children's Emotional States and Parental Anxiety. J Perianesth Nurs. 2018 Dec;33(6):972-980. doi: 10.1016/j.jopan.2017.09.008. Epub 2017 Nov 20. PMID 30449445
- [Result] 1. Atalay B, Güler R.,Haylı Ç.M.(2021). Investıgatıon Of Preoperatıve Anxıety Levels In Pedıatrıc Groups. Turkish Journal of Health Science and Life, 4(1); 24-26.
- [Result] Baghele A, Dave N, Dias R, Shah H. Effect of preoperative education on anxiety in children undergoing day-care surgery. Indian J Anaesth. 2019 Jul;63(7):565-570. doi: 10.4103/ija.IJA_37_19. PMID 31391620
- [Result] 4. Bülbül, F., &Arıkan B. (2018).Çocuklarda ameliyat öncesi psikolojik hazırlık:Güncel Yaklaşımlar. Balikesir Saglik Bil Derg 7(3).
- [Result] 5. Çelik S. (2020). Pediatrik triyajda palyaço uygulamasinin çocukebeveynin anksiyete ve memnuniyetine etkisi. İstanbul Üniversitesi-Cerrahpaşa Lisansüstü Eğitim Enstitüsü, Doktora tezi, 2021.
- [Result] Chartrand J, Tourigny J, MacCormick J. The effect of an educational pre-operative DVD on parents' and children's outcomes after a same-day surgery: a randomized controlled trial. J Adv Nurs. 2017 Mar;73(3):599-611. doi: 10.1111/jan.13161. Epub 2016 Oct 20. PMID 27681601
- [Result] Eijlers R, Dierckx B, Staals LM, Berghmans JM, van der Schroeff MP, Strabbing EM, Wijnen RMH, Hillegers MHJ, Legerstee JS, Utens EMWJ. Virtual reality exposure before elective day care surgery to reduce anxiety and pain in children: A randomised controlled trial. Eur J Anaesthesiol. 2019 Oct;36(10):728-737. doi: 10.1097/EJA.0000000000001059. PMID 31356373
- [Result] Getahun AB, Endalew NS, Mersha AT, Admass BA. Magnitude and Factors Associated with Preoperative Anxiety Among Pediatric Patients: Cross-Sectional Study. Pediatric Health Med Ther. 2020 Dec 16;11:485-494. doi: 10.2147/PHMT.S288077. eCollection 2020. PMID 33364873
- [Result] Moura LA, Dias IM, Pereira LV. Prevalence and factors associated with preoperative anxiety in children aged 5-12 years. Rev Lat Am Enfermagem. 2016 Jun 14;24:e2708. doi: 10.1590/1518-8345.0723.2708. PMID 27305179
- [Result] 10. Okyay R.D.,Ayoğlu H.(2018). Çocuklarda Postoperatif Ağrı Yönetimi. Pediatr Pract Res; 6(2):16-25.
- [Result] Binay Yaz S, Bal Yilmaz H. The Effects of Designing an Educational Animation Movie in Virtual Reality on Preoperative Fear and Postoperative Pain in Pediatric Patients: A Randomized Controlled Trial. J Perianesth Nurs. 2022 Jun;37(3):357-364. doi: 10.1016/j.jopan.2021.04.015. Epub 2022 Feb 15. PMID 35177320